CLINICAL TRIAL: NCT00892593
Title: Augmentation of Screening Colonoscopy With Fecal Immunochemical Testing
Acronym: ASC-FIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Forsyth Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ASC-FIT
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Colon Cancer
Keywords: colon; neoplasia; polyp; adenoma; FIT; cancer
MeSH Terms: conditions — Colonic Neoplasms; Neoplasms; Polyps; Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 Fecal Immunochemical Testing-Surveillance (Experimental): Fecal Immunochemical Testing performed at yearly intervals.
  Interventions: Device: Fecal Immunochemical Testing
- 2 Usual Care - Surveillance (No Intervention)
- 3 Usual Care - Screening (No Intervention)
- 4 Fecal Immunochemical Testing-Screening (Experimental): Fecal Immunochemical Testing yearly, beginning at year 6.
  Interventions: Device: Fecal Immunochemical Testing

INTERVENTIONS:
Device: Fecal Immunochemical Testing — Fecal Immunochemical Testing is a stool test specific for human hemoglobin.
  Other Names: FIT
  Arms: 1 Fecal Immunochemical Testing-Surveillance
Device: Fecal Immunochemical Testing — Fecal Immunochemical Testing is a stool test specific for human hemoglobin.
  Other Names: FIT
  Arms: 4 Fecal Immunochemical Testing-Screening

SUMMARY:
The study will determine if adding fecal immunochemical testing (FIT) at yearly intervals to a colonoscopy screening program will improve colon cancer detection rates.

DETAILED DESCRIPTION:
This study will evaluate the benefit of augmenting a compliant College of Gastroenterology colorectal cancer screening program with the addition of yearly FIT testing at two critical points in the current recommended follow up: 1. In patients found to have adenomatous polyps for the first time after colonoscopy, the addition of FIT in yearly intervals following index colonoscopy and 2. For subjects with "clean" colonoscopies (no polyps found), the addition of FIT at yearly intervals starting in year 6 and continuing to year 10 or subsequent colonoscopy. Current screening guidelines do not recommend the combination of colonoscopy and FOBT.

Two factors plague an effective colon cancer screening program: 1) a less than 100% sensitivity (95% ) for optical colonoscopy to detect colon cancer, and 2) Limitations of guaiac based stool testing: low sensitivity ( 5% in single use) for detection of colon cancer and the traditional gFOBT is cumbersome for patients to perform, impeding patient acceptance and adherence.

FIT offers a FOBT with improved sensitivity (65% for invasive colon cancer) and improved specificity and better patient compliance. The addition of FIT after initial colonoscopy could be applied to a screening program and thereby salvage "missed" lesions by increased detection rates

ELIGIBILITY:
Inclusion Criteria:

Group I (positive colonoscopy)

* 18 to 75 years of age
* male or female
* willing to provide written informed consent
* In the event that the colonoscopy is incomplete, or polypectomy is partial, the above patients are eligible if a successful examination is completed within 6 months of the inadequate exam.

Group II (negative colonoscopy)

* 50 to 69 years of age
* Male or female
* Willing to provide written informed consent
* In the event that the colonoscopy is incomplete, the patient is eligible if a successful examination is completed within 6 months of the inadequate exam.

Exclusion Criteria:

Group I (positive colonoscopy)

* chronic use of coumadin
* history of previous GI malignancy, inflammatory bowel disease (Crohns disease, ulcerative colitis)
* age or health status contraindicates repeat colonoscopy
* history of Familial Polyposis or Hereditary Nonpolyposis Colon Cancer Syndrome
* The index colonoscopy resulted in a perforation requiring surgical repair
* An otherwise qualifying colonoscopy is followed by a recommendation for repeat colonoscopy in ≤ 1 yr.

Group II (negative colonoscopy)

* chronic use of coumadin
* history of previous GI malignancy, inflammatory bowel disease (Crohns disease, ulcerative colitis)
* age or health status contraindicates repeat colonoscopy
* history of Familial Polyposis or Hereditary Nonpolyposis Colon Cancer Syndrome
* The index colonoscopy resulted in a perforation requiring surgical repair
* Significant family history resulting in a recommendation for repeat colonoscopy in 5 years or less

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4100 (Estimated)
Dates: Start 2009-05; Primary Completion 2019-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
rate of significant colon neoplasia among those who enter a screening or surveillance program with FIT testing added at yearly intervals vs. that of "usual care" patients in the same patient population. | yearly

SECONDARY OUTCOMES:
the pathology found at repeat colonoscopy in each group. | Yearly

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Murphy, M.D., Principal Investigator — Piedmont Gastroenterology Specialists
Locations (3):
- United States (3):
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - Piedmont Gastroenterology Specialists, PA, Winston-Salem, North Carolina
  - Salem Gastroenterology Associates, PA, Winston-Salem, North Carolina

REFERENCES:
- See also: NovantHealthClinicalResearch/ASC-FIT — http://www.novanthealth.org/forsyth-medical-center/services/clinical-research.aspx